CLINICAL TRIAL: NCT07209462
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of MRM-3379 in Male Participants With Fragile X Syndrome
Brief Title: Study of MRM-3379 in Male Participants With Fragile X Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENV-202
Record Dates: First submitted 2025-10-02; First posted 2025-10-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; FXS; FMR; Phosphodiesterase 4; PDE4
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: Low Dose of MRM-3379 (Experimental): Participants 16-45 years of age randomized to this arm will receive the low dose of MRM-3379
  Interventions: Drug: Low dose of MRM-3379
- Arm 2: Middle dose of MRM-3379 (Experimental): Participants 16-45 years of age randomized to this arm will receive the middle dose of MRM-3379
  Interventions: Drug: Middle Dose of MRM-3379
- Arm 3: High dose of MRM-3379 (Experimental): Participants 16-45 years of age randomized to this arm will receive the high dose of MRM-3379
  Interventions: Drug: High dose of MRM-3379
- Arm 4 :Placebo (Placebo Comparator): Participants 16-45 years of age randomized to this arm will receive Placebo
  Interventions: Drug: Placebo
- Arm 5: Low dose of MRM-3379 Open-Label (Experimental): Participants 13 to < 16 years of age will receive the low dose of MRM-3370 Open-Label
  Interventions: Drug: Low dose of MRM-3379 Open-Label

INTERVENTIONS:
Drug: Low dose of MRM-3379 — Oral capsule
  Arms: Arm 1: Low Dose of MRM-3379
Drug: Middle Dose of MRM-3379 — Oral capsule
  Arms: Arm 2: Middle dose of MRM-3379
Drug: High dose of MRM-3379 — Oral capsule
  Arms: Arm 3: High dose of MRM-3379
Drug: Placebo — Capsules matched to study drug without the active pharmaceutical ingredient
  Arms: Arm 4 :Placebo
Drug: Low dose of MRM-3379 Open-Label — Oral capsule
  Arms: Arm 5: Low dose of MRM-3379 Open-Label

SUMMARY:
This study is a multicenter, double-blind, randomized, placebo-controlled study to assess the safety and tolerability of 3 doses of MRM-3379 in male participants with Fragile X Syndrome ages 16 to 45 (inclusive). In addition, a parallel cohort of participants ages 13 to <16 will receive open-label MRM-3379. All participants will participate for 12 weeks of treatment. The study is also intended as a proof-of-concept investigation to evaluate whether MRM-3379 can improve FXS symptoms

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed informed consent/assent. Where local regulations permit inclusion of participants deemed unable to provide informed consent, a legally authorized representative must provide informed consent on the participant's behalf, and the participant must provide assent if applicable.
* Male, 13-45 years of age (inclusive)
* Weight ≥30 kg and BMI between 18 and 36 kg/m2 (inclusive) at the screening visit
* Diagnosis of FXS with a molecular genetic ≥200 CGG repetitions .
* Able to perform the PVT and ORRT of the NIH-TCB
* Have a consistent caregiver(s) who is willing and able to be present regularly and reliably with the participant
* Able to swallow tablets or capsules

Exclusion Criteria:

History of or current medical condition other than FXS and related issues that would place the participant at higher risk from study participation

Ages: 13 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 60 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events and Withdrawal due to adverse events and withdrawal due to adverse events | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Amnova Clinical Research, LLC, Irvine, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Suburban Research Associates, Media, Pennsylvania

IPD SHARING:
Plan to Share IPD: No